CLINICAL TRIAL: NCT03808779
Title: A Multicenter, Randomized and Controlled Trial of Radiofrequency Ablation vs. Conventional Surgery as Treatment of Papillary Thyroid Microcarcinoma (PTMC)
Brief Title: A Multicenter Trial of Radiofrequency Ablation vs. Surgery as Treatment of Papillary Thyroid Microcarcinoma.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, huang pintong, Director of Department of Ultrasound, Professor of Zhejiang University School of Medicine, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-004-A012
Record Dates: First submitted 2019-01-13; First posted 2019-01-18 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Papillary Thyroid Microcarcinoma
Keywords: Papillary Thyroid Microcarcinoma; Radiofrequency Ablation; Surgery
MeSH Terms: conditions — Papillary Thyroid Microcarcinoma | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency Ablation (Experimental): Eligible participants with PTMC will be randomly assigned to this group and undergo radiofrequency ablation(RFA) procedure.
  Interventions: Procedure: Radiofrequency Ablation
- Conventional Surgery (Active Comparator): Eligible participants with PTMC will be randomly assigned to this group and undergo total/thyroid lobectomy procedure.
  Interventions: Procedure: Conventional Surgery

INTERVENTIONS:
Procedure: Radiofrequency Ablation — Patients were supine with the neck exposure completely during the procedure. Local anesthesia with 1% lidocaine was injected at the subcutaneous puncture site and the thyroid anterior capsule. If the distance between the tumor and critical cervical structures was less than 5 mm, normal saline was injected to form at least 1 cm distance between the tumor and the critical structure to prevent the unwilling thermal injury. RFA was performed using the moving-shot technique and RFA power was 5 W, if a transient hyperechoic zone did not form at the electrode tip within 5-10 seconds. The RFA extent exceeded the tumor edge to prevent marginal residue and recurrence. The ablation was terminated when all portions of the target ablation area had changed to hyperechoic zones.
  Other Names: RFA
  Arms: Radiofrequency Ablation
Procedure: Conventional Surgery — Patient is performed total thyroidectomy or thyroid lobectomy depending on the intraoperative situation, disease condition and comprehensive judge by surgeon. Patients are routinely disinfected and spread the drapes after general anesthesia. Neck skin, fat and placenta muscle are incised and separated successively. The flap is separated to the upper edge of thyroid cartilage, neck white line is incised and anterior muscle group is separated. Then both sides thyroid lobes are exposed. Cut off the isthmus, ligature the thyroid artery, cut off the upper pole. Ligature and cut off the ipsilateral thyroid vein. Reveal and protect the ipsilateral recurrent laryngeal nerve and the parathyroid gland during the entire process.
  Other Names: Total thyroidectomy/Thyroid lobectomy
  Arms: Conventional Surgery

SUMMARY:
The treatment of Papillary Thyroid Microcarcinoma (PTMC) nowadays varies among physicians, surgeons and radiologist. The recently published articles show that the prognosis of PTMC by different means of treatment strategies tends to be good. But multicentered, randomized, parallel and prospective study is rare. RFA is the abbreviation of "Radiofrequency Ablation", which tends to be an alternative strategy except conventional surgery. The investigator aims to confirm whether RFA for treating PTMC braces same effectiveness and prognosis comparing with conventional surgery. Besides, this trial also investigates the safety, economy and psychological quality under different treatments.

DETAILED DESCRIPTION:
The incidence of thyroid carcinoma, especially the papillary thyroid microcarcinoma (PTMC), has increasingly rapidly, due to the development of technologies of diagnosis, during the past 20 years. PTMC defined by the World Health Organization (WTO) as the largest dimension less than 1 cm. Previous autopsy study demonstrated that the lesions are normal in many people and accompany them latently until they die because of another reasons. The long-term outcome of PTMC is good and, as expected, more than 90% PTMC aren't progress for many years.

Ultrasound-guided Radiofrequency Ablation (RFA) treatment was introduced to clinical practice few years ago. According to the 2015 American Thyroid Association (ATA) guideline, the treatment of radiofrequency and laser ablation are mentioned to be used in recurrent thyroid cancer. But clinical practice shows that the RFA treatment for low risk PTMC braces well effect，low financial budget，high safety and even rare postoperative complication.

Although the cohort study was performed before, the real answer concerning about whether RFA is a rational choice for treating PTMC lacks more powerful evidences. The investigator considers to perform a randomized, controlled and multicenter study as a high-quality evidence and demonstrated the effect of PRF in low risk PTMC treatment.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosis of PTMC (largest dimension<10mm)
* Age >=18 years old
* Bethesda Category V or VI
* Single nodule without thyroid capsule contact
* Nodule has more than 3mm distance far from recurrent laryngeal nerve, carotid artery and trachea.
* No clinical evidences show there is local or distant metastasis.
* Without chemotherapy, radiotherapy and other related therapies.
* Patients and their family member totally understand and sign the informed consent.

Exclusion Criteria:

* Multifocal PTMC
* Combined with other types of thyroid cancer or hyperthyroidism.
* Contralateral vocal cord paralysis
* With local or distant metastasis
* Pregnant woman
* With radiation exposure history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Recurrent-free Survival Rate | 5 years
  record detecting recurrence of PTMC post-surgery or post-FRA

SECONDARY OUTCOMES:
The Diameter of Lesion | 5 years
  record diameter reduce rate after RFA procedure
The Volume of Lesion | 5 years
  record volume reduce rate after RFA procedure
Postoperative Complications | up to 12 months
  record relevant complications after surgery or RFA
Serum Concentration of Serological Examination of Thyroid Function | up to 12 months
  record the serum concentration of TSH/T3/FT3/T4/FT4/TPOAb/TgAb/TRAb.
Medical Cost | up to 12 months
  record hospital expenditure
Hospital Duration | through study completion, an average of 7 days
  record hospital stay time
Patient Satisfaction: questionnaire | 5 years
  measured by satisfaction questionnaire designed by investigator group： items：
  1．Are you satisfied with surgery? 2.Are you satisfied with the RFA procedure? scale range from 1 to 10； by the increasing of scale, the outcome is defined as good.
Anxiety index measured by psychological questionnaire | up to 5 years
  1. I feel more nervous and anxious than usual (anxiety)
  2. I feel scared for no reason (fear)
  3. I am easily upset or frightened (frightened)
  4. I think I might be going crazy (madness) There are 20 questions (No. 5-20 don't show because of the 999 words restriction).
  scale range from 1 to 4 For the question 5,9,13,17,18, the outcome is define as good by the increasing of scale.
  For the others, the outcome is defined as bad by the increasting of scale.(scale 1=No or very few, scale2=sometimes, scale3=often, scale4=always)
Overall Survival in Patients with PTMC | 5 years
  record 5 year overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Pintong Huang, director, Principal Investigator — Department of Ultrasound, Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (3):
- China (2):
  - General Surgery Department, Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Department of Ultrasound, Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
- Interventional Oncology Centre, State Institution "Grigoriev Intstitute for Medical Radiology NAMS of Ukraine", Kharkiv, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided